CLINICAL TRIAL: NCT00405470
Title: A Prospective Randomized Trial Using Roentgen Stereophotogrammetric Analysis of the Advance Medial Pivot Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Michael Gross, MD FRCSC PhD, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAL06-01
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Osteoarthritis, Knee
Keywords: arthroplasty; RSA; micromotion; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medial Pivot (Active Comparator)
  Interventions: Device: Advance Medial Pivot Knee Arthroplasty
- Posterior Stabilized (Active Comparator)
  Interventions: Device: Advance Medial Pivot Knee Arthroplasty

INTERVENTIONS:
Device: Advance Medial Pivot Knee Arthroplasty — medial pivot total knee arthroplasty tibial component vs standard posterior stabilized tibial component with post. Medial pivot provides a constrained medial condyle through shape of polyethylene and reduces amount of bone removal on femoral side that would otherwise be removed to accommodate PS post

SUMMARY:
The purpose of this study is to determine whether this particular knee replacement is better than those already on the market. By participation, it will further refine the design of future total knee replacements and perhaps increase longevity.

DETAILED DESCRIPTION:
Joint arthroplasty is an effective surgical intervention, however prosthetic survivorship is finite. New or modified prosthetic components are routinely introduced, partly in an effort to improve survivorship. When new technologies emerge for total knee replacement it is not always evident that they are an improvement over existing options. This determination requires long-term follow-up studies. Conventional studies require a large number of patients and approximately 10 years of follow-up. By using RSA to measure micromotion of prostheses over time problems can be elucidated with a much smaller sample over a shorter time period. RSA involves using tantalum markers (0.5-1.0 mm beads inserted in the bone and prosthesis during surgery) to measure motion in subsequent bi-planar x-rays of the joint. The relatively new Medial Pivot Knee (ADVANCE Knee) theoretically reproduces the natural kinematics of the knee but it is unclear what effect this design may have on the forces applied to the tibial component-bone interface. The amount of micromotion of the tibial component is directly related to the amount of force exerted on it and inversely related to its fixation. In this study we propose to compare in vivo micromotion at the tibial component-bone interface with the ADVANCE Medial-Pivot Knee (experimental group) versus a more conventional prosthesis (control), the ADVANCE Traditional Knee. Patients (n=60; age 45-80 years old) with primary osteoarthritis of the knee and mono-articular disease will be randomized to receive either the ADVANCE Traditional or ADVANCE Medial-Pivot Knee using Simplex cement. Eight tantalum markers will be placed in both the tibia and femur proximal to the prosthesis and in the polyethylene tray of the tibial component. Pre-operatively and at 6, 12 and 24 months all patients will complete general health (SF-12) and joint specific questionnaires (Oxford -12 Item Knee Score), have their body mass index calculated, and have the range of motion, alignment, extensor function and ligamentous competency of their index knee recorded. On the first weight-bearing day after surgery bi-planar standing x-rays will be taken and used as a reference point for tibial component position. At 6, 12 and 24 months post-operatively patients will undergo more bi-planar standing x-rays incorporating provocative loading tests. Micromotion will be analyzed through serial comparison of digital x-rays by blinded study personnel using RSA software. Parametric statistics (unpaired Student's t-test) will be used to compare the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee
* Mono-articular disease (Charnley Modified Type A)

Exclusion Criteria:

* Significant co-morbidity affecting ability to ambulate
* Flexion contracture greater than 15°
* Tibial subluxation greater than 10 mm on standing AP radiograph
* Greater than 10° of varus or 15° of valgus
* Extension lag greater than 10°
* Lateral or medial collateral ligament instability (> 10° varus/valgus)
* Previous osteotomy about the knee
* Previous arthroplasty of the knee
* Previous patellectomy
* Leg length discrepancy greater than 10 mm
* Morbid obesity (obesity that results in significant systemic problems)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-07; Primary Completion 2005-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
tibial implant micromotion relative to tibia at 2 years | 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gross, MD FRCSC PhD, Principal Investigator — Dalhousie University & Capital District Health Authority